CLINICAL TRIAL: NCT03727880
Title: A Randomized Phase II Study of Pembrolizumab With or Without Defactinib, a Focal Adhesion Kinase Inhibitor Following Chemotherapy as a Neoadjuvant and Adjuvant Treatment for Resectable Pancreatic Ductal Adenocarcinoma (PDAC)
Brief Title: Study of Pembrolizumab With or Without Defactinib Following Chemotherapy as a Neoadjuvant and Adjuvant Treatment for Resectable Pancreatic Ductal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lei Zheng (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Verastem, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Lei Zheng, Executive Director of University of Texas Health Science Center at San Antonio Cancer Center, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTMS 25-0012; STUDY00001506 (Other: UTHSCSA IRB)
Record Dates: First submitted 2018-10-31; First posted 2018-11-01 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Resectable Pancreatic Ductal Adenocarcinoma (PDAC); Pancreatic Ductal Adenocarcinoma
Keywords: Pembrolizumab; Defactinib; Immunotherapy; Anti-PD-1; Antibody; PD-L1; Pancreatic cancer; Neoadjuvant chemotherapy; Adjuvant chemotherapy; PDAC - Pancreatic Ductal Adenocarcinoma; FAK (focal adhesion kinase) inhibitor; Resectable Pancreatic Adenocarcinoma; High Risk Resectable Pancreatic Cancer; Tumor microenvironment; CA 19-9; Surgery; Pancreatectomy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pembrolizumab; defactinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - Pembrolizumab and Defactinib (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: Defactinib
- Arm B - Pembrolizumab (Experimental)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Following standard of care neoadjuvant chemotherapy, subjects will receive two doses of pembrolizumab (200mg) IV 3 weeks apart prior to surgery. After surgery, subjects will receive adjuvant standard of care chemotherapy. Following adjuvant chemotherapy, subjects will receive 8 doses of pembrolizumab (200mg) IV 3 weeks apart.
  Other Names: MK-3475; Keytruda
Drug: Defactinib — Following 2 cycles of standard of care neoadjuvant chemotherapy, subjects will receive 400 mg defactinib twice a day up until 2 days preceding their surgery (approximately 6 weeks) during the immunotherapy cycles with pembrolizumab. After surgery, subjects will receive adjuvant standard of care chemotherapy. Following adjuvant chemotherapy, subjects will receive 400mg defactinib twice a day for 24 weeks.
  Arms: Arm A - Pembrolizumab and Defactinib

SUMMARY:
This study will test the effectiveness (anti-tumor activity), safety, and ability to increase the body's immune system to fight pancreatic cancer by combining standard chemotherapy before and after surgery, with study drug PD-1 antibody, pembrolizumab, with and without study drug, focal adhesion kinase inhibitor (FAK), defactinib, in people with "high risk" resectable (surgically removable) pancreatic cancer. The purpose of this study is to evaluate if reprograming the tumor microenvironment by targeting FAK following chemotherapy can potentiate anti-programmed death-1 (PD-1) antibody.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Has pancreatic ductal adenocarcinoma
* Has resectable disease at the time of diagnosis
* Has not received any systemic therapy for pancreatic ductal adenocarcinoma
* Has stage ≤ IIb disease at time of diagnosis and enrollment
* Elevated tumor marker, CA (carbohydrate antigen) 19-9 >200
* ECOG performance status 0 or 1
* Patient must have adequate organ function defined by the study-specified laboratory tests.
* Must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

Patients who have received any prior chemotherapy, radiotherapy or investigational agents for pancreatic cancer.

* Patients who have received prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).
* Has received prior therapy with FAK inhibitor.
* Woman who are pregnant or breastfeeding.
* Have received a live vaccine or live-attenuated vaccine within 30 days prior to study drug.
* Is currently or has participated in another investigational study within 4 weeks prior to receiving study drug.
* History or current use of immunosuppressive medications within 7 days prior to study medications.
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years or that is expected to require active treatment within two years.
* Has active autoimmune disease that has required systemic treatment in the past 2 years.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Infection with HIV or hepatitis B or C.
* Patient with uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known allergy or hypersensitivity to the study drugs.
* Received any growth factors including, but not limited to, granulocyte-colony stimulating factor (G-CSF), GM-CSF, erythropoietin, within 14 days of study drug administration.
* Has history of any organ transplant, including corneal transplants.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zheng, MD, Principal Investigator — The University of Texas Health Science Center San Antonio; Arsen Osipov, MD, Study Chair — Cedar Sinai
Locations (3):
- United States (3):
  - Samuel Oschin Cancer Center at Cedars-Sinai, Los Angeles, California
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - The University of Texas Health Science Center San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fard D, Giraudo E, Tamagnone L. Mind the (guidance) signals! Translational relevance of semaphorins, plexins, and neuropilins in pancreatic cancer. Trends Mol Med. 2023 Oct;29(10):817-829. doi: 10.1016/j.molmed.2023.07.009. Epub 2023 Aug 17. PMID 37598000

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A - Pembrolizumab and Defactinib | Arm B - Pembrolizumab
Started | 14 | 14
Completed | 13 | 10
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Population: Number of evaluable participants randomized to interventions
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Pembrolizumab and Defactinib | Arm B - Pembrolizumab | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.54 (11.39) | 73.5 (6.62) | 72.4 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR) Rate
Description: Percent of subjects with a pathologic complete response (pCR) per the tumor regression grade scores established by the College of American Pathologist: Grade 0= complete response (no viable cancer cells), Grade 1= near complete response (single cells or rare small groups of cancer cells), Grade 2= partial response (residual tumor with evidence of regression), or Grade 3= no response (extensive residual tumor with no evidence of regression).
Time Frame: 4 years
Population: Participants that reached pCR
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A - Pembrolizumab and Defactinib | Arm B - Pembrolizumab
Number analyzed (Participants) | 10 | 8
Percentage of participants | 0 | 0

2. Secondary Outcome: Overall Survival (OS)
Description: Number of months until death
Time Frame: 4 years
Population: Participants evaluable were those that were randomized to intervention and completed the study
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Arm A - Pembrolizumab and Defactinib | Arm B - Pembrolizumab
Number analyzed (Participants) | 13 | 10
months | 25.01 (14.48) | 27.39 (19.54)

3. Secondary Outcome: Disease Free Survival (DFS)
Description: Number of months until disease recurrence
Time Frame: 4 years
Population: For Arm A overall study was completed by 13 pt, DFS evalauted for 11. The remaining 2 participants were not evaluable for DFS because surgery was not performed and therefore they never achieved a disease-free baseline For Arm B overall study was completed by 10 pt, DFS evalauted for 8. The 2 participants whose surgeries were attempted but aborted were not evaluable for DFS because they never achieved a disease-free baseline."
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Arm A - Pembrolizumab and Defactinib | Arm B - Pembrolizumab
Number analyzed (Participants) | 11 | 8
months | 16.59 (14.33) | 15.99 (15.20)

4. Secondary Outcome: Number of Participants Experiencing Study Drug-related Toxicities
Description: Number of participants experiencing drug-related adverse events as defined by CTCAE v5.0
Time Frame: 4 years
Population: Includes all participants that both completed and did not complete the study
Measure: Number; unit: participants
Arm/Group | Arm A - Pembrolizumab and Defactinib | Arm B - Pembrolizumab
Number analyzed (Participants) | 14 | 14
participants | 6 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to 4 years
Description: Adverse events were assessed according to CTCAEv5.0
Arm/Group | Arm A - Pembrolizumab and Defactinib | Arm B - Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 10/14 | 6/14
Serious Adverse Events (participants affected / at risk) | 2/14 | 3/14
Other Adverse Events (participants affected / at risk) | 4/14 | 3/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Pembrolizumab and Defactinib (N=14) | Arm B - Pembrolizumab (N=14)
Non-pancreatic cancer (General disorders) | 2 (2) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Pembrolizumab and Defactinib (N=14) | Arm B - Pembrolizumab (N=14)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (8)
Increased bilirubin (Blood and lymphatic system disorders) | 3 (9) | 0 (0)
Elevated aspartate aminotransferase (AST) (Hepatobiliary disorders) | 1 (7) | 0 (0)
Elevated Alanine transaminase (ALT) (Hepatobiliary disorders) | 1 (8) | 0 (0)
Acnieform rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT03727880/Prot_SAP_000.pdf